CLINICAL TRIAL: NCT02458950
Title: Characteristics and Clinical Outcomes of Anorexia Nervosa : Siriraj Hospital Experience
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: Si501/2014
Record Dates: First submitted 2015-05-28; First posted 2015-06-01 (Estimated); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia nervosa; Siriraj Hospital; Thai
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is aimed to determine clinical characteristics of patients with anorexia nervosa and outcome of treatment at Sirirraj Hospital.

DETAILED DESCRIPTION:
Data is derived from the medical records

ELIGIBILITY:
Inclusion Criteria:

* children and adolescents with newly diagnosed anorexia nervosa in Siriraj Hospiatl according to DSM IV criteria
* treated by multidisciplinary teams e.g. pediatricians specialized in nutrition and psychology and psychologist

Exclusion Criteria:

* none

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients of Siriraj Hospital
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
types and factors contributing to outcomes of anorexia nervosa | one year

SECONDARY OUTCOMES:
Outcome of treatment of anorexia nervosa | one year
  By using core symptoms (bodyweight, menstruation, and eating behavior), outcome can be categorized into 4 groups, which are recovery, improvement, chronicity, and death.

CONTACTS AND LOCATIONS:
Overall Officials: Narumon Densupsoontorn, MD, Study Chair — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand

REFERENCES:
- [Background] Nakai Y, Nin K, Noma S, Hamagaki S, Takagi R, Wonderlich SA. Outcome of eating disorders in a Japanese sample: a 4- to 9-year follow-up study. Eur Eat Disord Rev. 2014 May;22(3):206-11. doi: 10.1002/erv.2290. Epub 2014 Mar 14. PMID 24634188
- [Result] Goldstein MA, Dechant EJ, Beresin EV. Eating disorders. Pediatr Rev. 2011 Dec;32(12):508-21. doi: 10.1542/pir.32-12-508. No abstract available. PMID 22135421